CLINICAL TRIAL: NCT05460858
Title: Effect of N-acetyl Cysteine on Oxidative Stress Biochemical Factors and IVF/ICSI Outcomes in Women With Endometrioma: A Randomized, Double-blinded, Phase III Clinical Trial
Brief Title: NAC Effect on Infertile Women With Endometrioma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Royan-NAC-Genetics
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Female Infertility; Endometrioma; Stress Oxidative
Keywords: en
MeSH Terms: conditions — Infertility, Female; Endometriosis | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-acetyl cystein (Experimental): Seventy participants who randomly assigned in the intervention group, during 6 weeks simultaneous to start standard long agonist protocol or antagonist induction, will be received 1200 (2×600) mg of effervescent tablets of NAC daily. Plasma blood will collect before the intervention and at the time of oocyte retrieval (end of 6 week), in addition to, follicular fluid will be obtained from the mature follicles. Also, we will measure severity of dysmenorea by visual analogue scale (VAS) technique.
  Interventions: Drug: N-acetyl cysteine
- effervescent placebo (Placebo Comparator): Seventy participants who randomly assigned to the control group, during 6 weeks simultaneous to start the standard long agonist protocol, or antagonist induction, will be received 1200 (2×600) mg of effervescent placebo tablets daily. Plasma blood will collect before the intervention and at the time of oocyte retrieval, in addition to, follicular fluid will be obtained from the mature follicles. Also, we measure severity of dysmenorrhea by visual analogue scale (VAS) technique.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: N-acetyl cysteine — One hundred and forty participants randomize in the intervention and placebo groups, during 6 weeks simultaneous to start standard long agonist protocol or antagonist induction. They will be received 1200 (2×600) mg of effervescent tablets of NAC or placebo daily. Plasma blood will collect before the intervention and at the time of oocyte retrieval (end of 6 week), in addition to, follicular fluid will be obtained from the mature follicles.
  Arms: N-acetyl cystein
Drug: placebo — placebo
  Arms: effervescent placebo

SUMMARY:
Oxidative stress has been investigated as a key factor in the pathogenesis and progression of endometrioma. High follicular fluid ROS levels and serum can be related to negative IVF/ICSI outcomes in infertile women with endometrioma. Therefore, the use of antioxidants such as N-acetyl cysteine (NAC) may be reduced complications of endometrioma. To study this hypothesis, we designed a double-blind, randomized clinical trial study that aimed to determine the effect of N-acetyl cysteine (NAC) on stress oxidative factors and pregnancy outcomes in IVF/ICSI cycles in endometrioma patients.

DETAILED DESCRIPTION:
This study will be conducted at Royan institute on 140 women with endometrioma who are eligible for the study after receiving written consent. After randomization, the participants will be divided into two intervention and control groups. Then, they will be received 1200 (2×600) mg of effervescent tablets of NAC or the placebo daily during 6 weeks simultaneous to start standard long agonist or antagonist protocols for induction.

Plasma blood will be collect before intervention and at the time of egg retrieval, in addition to, follicular fluid (FF) will be obtained from the mature follicles of each ovary and will be separated by centrifuging and will be frozen until analysis. Then, we will measure the levels of two markers of oxidative stress (TAC: Total antioxidant capacity and SOD: Superoxide dismutase) in plasma and FF of all samples by enzyme-linked immunosorbent assay (ELISA) method. In addition, the pregnancy outcomes will be investigated in treated and untreated groups. Also, we will study the effect of pain severity of by visual analogue scale (VAS) technique.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 42 years
* Ultrasound or laparoscopic diagnosis of moderate to sever endometrioma (endometriosis stage III and IV)
* Serum AMH levels between 0.7 and 4.5 ng/ml
* Standard long GnRH and antagonist ovulation stimulation cycle
* Body mass index (BMI) <30 kg/m2

Exclusion Criteria:

* Non-inclusion criteria: Congenital uterine malformations
* Severe male infertility (TESE, PESA)
* Past medical history of asthma

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2023-09-23 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
MII oocyte number and quality | Immediately after oocyte puncture
  Observation of oocytes that were mature at the time of oocyte collection

SECONDARY OUTCOMES:
Measurement of TAC oxidative stress marker in blood plasma | Before intervention and 6 weeks after intervention
  Plasma will be obtained for studying TAC and measure by ELISA
Measurement of SOD oxidative stress marker in blood plasma | Baseline and 6 weeks after intervention
  Plasma will be obtained for studying SOD and measure by ELISA
Measurement of TAC oxidative stress marker in folicular fluid | Immediately After oocyte puncture
  Folicular fluid will be obtained for studying TAC and measure by ELISA
Measurement of SOD oxidative stress marker in folicular fluid | Immediately After oocyte puncture
  Folicular fluid will be obtained for studying SOD and measure by ELISA
Cleaved embryo numbers | 2-3 days after oocyte puncture
  2-3 days embryo from fertilization
Blastocyst numbers | 5 days after oocyte puncture and sperm insemination
  The stage the embryo reaches after 5 days in culture from the egg retrieval
Clinical pregnancy rate | 4-6 weeks after embryo transfer
  The observation of gestational sac on ultrasound examination two-three weeks after positive serum βhCG
Fertilization rate | 2-5 days after sperm insemination
  Percentage of transformation of micro injected oocytes into two pronuclei embryo

CONTACTS AND LOCATIONS:
Overall Officials: Parvaneh Afsharian, PhD, Principal Investigator — Royan Institute
Locations (1):
- Royan Institute, Tehran, Iran